CLINICAL TRIAL: NCT05294133
Title: Implementation of a 12-week Adapted Physical Activity (APA) Program in People Suffering From Chronic Insomnia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-A00862-39
Record Dates: First submitted 2021-12-10; First posted 2022-03-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Exercise; Health Behavior; Sleep
MeSH Terms: conditions — Motor Activity; Health Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention
- physical activity (Experimental)
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — physical activity
  Arms: physical activity

SUMMARY:
One third of men and women are not satisfied with their sleep. A non-drug countermeasure to improve sleep in insomniacs could be adapted physical activity (APA). However, research is needed because the literature is limited and the few studies are most often based on subjective data with a great methodological disparity. Within the framework of the care pathway of Dr ARON's patients, sleep doctor at the Sommeil Morphée Center of the Grande Synthe Polyclinic (59), the objective of this project is to make an APA program more reliable in order to improve sleep, to understand the underlying mechanisms and to include APA in the therapeutic management.

DETAILED DESCRIPTION:
According to the 2019 National Sleep and Vigilance Institute survey, in France, one-third of men and women are not satisfied with their sleep, and nearly half struggle to fall asleep or return to sleep. Given the growing evidence of the harmful effects of lack of sleep, its alteration on health, these figures are alarming.

Insomnia is characterized by dissatisfaction with the quantity or quality of sleep, difficulty initiating and/or maintaining sleep, and early morning awakenings at least three times a week for a minimum period of three months.

In a Sleep Medicine Reviews report, it was shown that many patients diagnosed with insomnia had a physiological hyperarousal disorder that resulted in poor sleep, which has been found in insomniacs in numerous studies. It is observed in particular on the autonomic nervous system by a low variability of heart rate and a high level of noradrenaline reflecting a dominant sympathetic axis. An anxiogenic and depressive profile and elevated cortisol levels are also often associated with this hyperarousal encountered in insomniacs. In addition, an alteration of the circadian rhythm seems to favor insomnia. Indeed, a decrease in core temperature and cortisol levels in the evening are primary mechanisms for sleep onset. A study showed an elevated sleep latency in individuals with this delayed circadian temperature rhythm. In the same study, a high wake-up time after sleep was associated with a high core temperature. Regarding cortisol, a smaller decline in cortisol and higher cortisol levels at the end of the day are associated with shorter sleep duration, lower sleep efficiency, and poor subjective sleep quality.

Although a first treatment of insomnia would be to find a good lifestyle and optimal sleep conditions, the majority of first-line remedies in the treatment of insomnia remain pharmacological today, through the short- or medium-term prescription of hypnotics, neuroleptics, anxiolytic benzodiazepines or some antidepressants.

If the practice of regular physical activity is now well known to improve overall health, what about sleep?

In 2017, the investigators published a study showing that an adapted Physical Activity (PA) program improved sleep in a population of young women. Overall, studies regarding the effects of exercise and physical activity are still recent but increasingly confirm the beneficial effects of PA on sleep.

Indeed, the literature reveals that there is an inverse correlation between the amount of PA and the severity of sleep disturbance.

In fact, it appears that regular physical activity decreases the recurrence of insomnia. In adults over 40 years of age with sleep disorders, a 10- to 16-week training program very significantly improved the qualitý of sleep and shortened sleep latency.

According to these same authors, PA thus poses as a reliable alternative to pharmacological management by showing a positive effect of PA on sleep.

However, further work is needed because the literature remains limited and sometimes contradictory. Moreover, the studies are most often based on subjective data with a great methodological disparity. The type of physical activity proposed in these different studies is very variable, ranging from aerobic exercise to muscle strengthening to yoga or other relaxation activities. To the best of our knowledge, there is no consensus on the intensity of exercise to be preferred to improve sleep.

1.1 Objectives

The objective of this project is therefore to evaluate the effects of an APA program in insomnia treatment therapies.

The follow-up of physiological and medical markers, throughout the APA program, will make it possible to observe the effect of the DK pulse intervention, to determine the mechanisms underlying the improvement of sleep by physical activity and thus to propose an optimization of the programs dedicated to the improvement of sleep.

The aim will be to extend this program from the local basin to the regional level (or even beyond) and to use the network of local APA structures to make this management as easy as possible for the patients.

1.1 General assumptions

The investigators hypothesize that the 12-week physical activity program will improve objective and subjective sleep in patients with insomnia. This improvement in sleep will be explained in part by a decrease in capillary cortisol levels, an increase in heart rate variability, a decrease in stress and/or an increase in circadian rhythm amplitude throughout the PA program.

This study is the second of three studies of the thesis of Pauline Baron (ULCO PhD student, financed by the Haut de France Region, in collaboration with health care services (Dr Aron).

The treating physicians of patients suffering from insomnia direct their patients to the dedicated sleep consultations for clinical assessment.

The sleep specialists propose physical activity within the framework of a prescription, after diagnostic and etiological assessments, and evaluation of the patients' symptoms, the comorbidities are evaluated in the same way as the motivation of the participants, and they ask the patients grouping the various criteria of inclusion/exclusion of the study if they wish to participate in a scientific study.

After the patient's informed consent, they are referred to Pauline BARON.

During the inclusion visit, the investigator reminds them in detail of the objectives and the course of the protocol. An information leaflet is given to each participant, who signs an authorization to participate in the study, accepting in particular the randomization of the groups (AP or control). The control group will not receive any intervention.

Adapted Physical Activities are programmed within the DK Pulse association, one of the 138 structures labelled Maison du Sport Santé (https://www.sports.gouv.fr/accueil-du-site/actualites/article/les-premieres-maisons-sport-sante-sont-desormais-connues ). The physical activity program is a 12-week program with 1 hour of aerobic type physical activity, of moderate intensity, 3 times a week (duration, frequency and intensity presumed to date according to the state of the art). The intensity of the physical activity (between 60 and 80% of VO2max) will be controlled by an RPE scale and a heart rate monitor.

The physical activity of the patients will be financially supported by the university.

As part of the care pathway, the investigators will evaluate different variables.

The variables will be measured at T0, T6 and T12 weeks for the 2 groups.

The following anthropometric and physiological parameters are measured:

Height (Tanita Leicester HR001 electronic height gauge); Body mass and composition (Tanita DC-360) Resting blood pressure (non-dominant arm, sitting position, Omron M3); White blood cell count measurement by capillary measurement (HemoCue® WBC DIFF Analyzer). Lack of sleep negatively affects the immune system. It is therefore interesting, especially in this health context, to measure the white blood cell count in patients suffering from insomnia, in order to prevent a possible infection.

Hair sampling for cortisol measurement (only at T0 and T12). The measurement of hair cortisol is essential in the care of a patient suffering from insomnia. It reflects the activity of the hypothalamic-pituitary-adrenal axis (HPA). An abnormally high level of cortisol and a disturbance of this axis can be a triggering or aggravating factor of insomnia.

Cardiorespiratory capacity on an ergometer (Monark e939): YMCA incremental submaximal test, up to 85% of the theoretical HR max, allowing to evaluate by projection the Maximum Aerobic Power (MAP) and the associated maximal O2 consumption (VO2max).

The evaluation is completed by taking an "e-celsius bodycap" capsule. This capsule allows continuous monitoring of the patient's core temperature. It is naturally eliminated in the stool. The follow-up of the central temperature is essential in the course of care of an insomniac patient. Indeed, it is one of the reflections of the biological clock and therefore allows us to observe the circadian rhythm and its amplitude.

At the end of this visit, patients will leave with :

an accelerometer, a Dreem research 2 headband a sleep diary and a physical activity log, a heart rate monitor (Polar H10).

During the following week, the participants equipped with the accelerometer on their wrist (non-dominant arm), fill out a daily sleep diary: wake-up and bedtime, naps.

They sleep with an EEG headband (Dreem 2 Research) that provides data for estimating the different stages of sleep.

The accelerometer allows to measure some sleep parameters such as total sleep time and time of nocturnal awakenings, the amount of physical activity and the associated energy expenditure (Actilife 6 software) during the 7 days. A PA diary will also be completed daily (type, intensity, duration).

Participants will wear the heart rate belt for 3 nights (from bedtime to sunrise) to record RR intervals (precise duration between each heartbeat) from which heart rate variability will be extracted (over a minimum interval of 5 hours). The frequency analysis of the RR signal allows to evaluate the respective activations of the sympathetic and parasympathetic nervous systems.

Each device is pre-programmed, no additional manipulation is necessary.

At the end of the 7 days, the participants return the equipment and answer several questionnaires:

On sleep and sleepiness: Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI) and EPWORTH sleepiness scale On stress and quality of life: Perceived Stress Scale (PSS) and the Short Form Health Study (SF 36) On PA level: International Fitness Scale (IFIS)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 60 with chronic insomnia (according to the 5 criteria of the Diagnostic and Statistical Manual) without any other associated sleep pathology (sleep apnea, restless legs syndrome, etc.)

Exclusion Criteria:

* Medical contraindication to physical activity Associated serious medical pathologies (cancer...) Night work, jet lag during the last month, young children BMI> 30 Current use or <3 months of psychoactive, hypnotic, stimulant or analgesic medications Alcohol or drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
subjective sleep change | before and after the 12 weeks
  questionnaire insomnia severity index. The minimum score is 0 and the maximum is 28. Higher scores mean a worse outcome. A score higher than 14 is considered as a person with clinical insomnia.
objective sleep change | before and after the 12 weeks
  Participants were fitted with an accelerometer on their wrist (non-dominant arm) for 7 days to assess the quantity and quality of their sleep

SECONDARY OUTCOMES:
circadian rythm change | before and after the 12 weeks
  continuous temperature with BodyCap capsules
objective stress change | before and after the 12 weeks
  cortisol level in hair
hearth rate variability change | before and after the 12 weeks
physical capacity change | before and after the 12 weeks
  Young Men's Christian Association (YMCA) submaximal VO2 test
subjective stress change | before and after the 12 weeks
  Perceived Stress Scale- 10. The minimum score is 10 and the maximum is 50. Higher scores mean a worse outcome. A score higher than 27 is considered as a person with very high perceived stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of littoral cote d'ople, Dunkirk, France

IPD SHARING:
Plan to Share IPD: No